CLINICAL TRIAL: NCT01795664
Title: A Double Blind, Double Dummy, Randomized, Two Way Cross-over Study to Compare the Effects of Seretide® Evohaler (Supplied by Allen & Hanburys, UK) and a Generic Salmeterol/Fluticasone HFA pMDI (Manufactured by Cipla Ltd, India) on Functional Respiratory Imaging Parameters in Asthmatic Patients.
Brief Title: Compare the Effects of Seretide® Evohaler and a Generic Salmeterol/Fluticasone Hydrofluoroalkane (HFA) Pressurized Metered-dose Inhaler (pMDI) on Functional Respiratory Imaging Parameters in Asthmatic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: FLUIDDA nv (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FLUI-2012-94; 2012-005789-36 (EudraCT Number); E-RES/12/12-Q13 (Other: Cipla Ltd, India)
Record Dates: First submitted 2013-01-31; First posted 2013-02-21 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Asthma
Keywords: Asthma; Salmeterol xinafoate and Fluticasone propionate; Seretide Evohaler; Functional Respiratory Imaging; Computational Fluid Dynamic
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Seretide Evohaler (Active Comparator): Salmeterol xinafoate and Fluticasone propionate combination HFA pMDI (Seretide Evohaler, Allen & Hanburys, UK)
  Strength: 25/250 mcg per actuation; Dose: single dose of 2 puffs; a total dose of 50/500 mcg
  Interventions: Radiation: Functional Respiratory Imaging; Drug: Seretide Evohaler; Drug: Placebo of Test product
- Salmeterol xinafoate and Fluticasone propionate HFA pMDI (Experimental): Salmeterol xinafoate and Fluticasone propionate combination HFA pMDI (Cipla Ltd., India)
  Strength: 25/250 mcg per actuation; Dose: single dose of 2 puffs; a total dose of 50/500 mcg
  Interventions: Radiation: Functional Respiratory Imaging; Drug: Salmeterol xinafoate and Fluticasone propionate HFA pMDI; Drug: Placebo of Reference product

INTERVENTIONS:
Radiation: Functional Respiratory Imaging — CT-scan of thorax, at visit 2 pre and postdose and at visit 3 pre and postdose
Drug: Salmeterol xinafoate and Fluticasone propionate HFA pMDI — Strength: 25/250 mcg per actuation; Dose: single dose of 2 puffs; A total dose of 50/500 mcg
  At visit 2 or visit 3 (cross-over design)
  Other Names: Test product
  Arms: Salmeterol xinafoate and Fluticasone propionate HFA pMDI
Drug: Seretide Evohaler — Strength: 25/250 mcg per actuation; Dose: single dose of 2 puffs; A total dose of 50/500 mcg
  At visit 2 or visit 3 (cross-over design)
  Other Names: Reference product; Salmeterol xinafoate and Fluticasone propionate combination HFA pMDI
  Arms: Seretide Evohaler
Drug: Placebo of Test product — Single dose of 2 puffs
  To ensure blinding, each patient will receive two inhalers (one active and one placebo) on each dosing day.
  Other Names: Placebo inhaler containing HFA propellant resembling the test active inhaler
  Arms: Seretide Evohaler
Drug: Placebo of Reference product — Single dose of 2 puffs
  To ensure blinding, each patient will receive two inhalers (one active and one placebo) on each dosing day.
  Other Names: Placebo inhaler containing HFA propellant resembling the reference active inhaler
  Arms: Salmeterol xinafoate and Fluticasone propionate HFA pMDI

SUMMARY:
This study will be conducted as a randomized, double blind, double dummy two period crossover study in stable asthma patients. A total of 16 stable asthma patients treated in accordance with the Global Initiative for Asthma (GINA) guidelines, will be included.

Objectives:

* The primary objective of this study is to evaluate the effect of both the study drugs under investigation on Functional Respiratory Imaging (FRI) parameters and to evaluate the particle deposition in the lungs using Computational Fluid Dynamic (CFD)
* The secondary objectives are to assess the effect of both the study drugs on lung function (spirometry and body plethysmography), on exercise capacity (6 Minutes Walking Test = 6MWT) and on dyspnea (Borg Category (C) Ratio (R) 10 Scale and Visual Analog Scale (VAS) dyspnea). Furthermore the safety of the 2 products under investigation will be evaluated through monitoring of adverse events (AEs) throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥ 18 years old
* Written informed consent obtained
* Patient with a documented diagnosis of asthma according to the GINA guidelines
* Patient with a co-operative attitude and ability to be trained to correctly use the pMDI
* Female patient of childbearing potential who confirm that a contraception method was used at least 14 days before visit 1 and will continue to use a contraception method during the study
* Patient must be stable and treated in accordance with the GINA guidelines
* Patient must be a non-smoker or ex-smoker who have stopped smoking at least 1 year prior to visit 1 and has a smoking history of < 10 pack years
* Patient must be able to understand and complete the protocol requirements, instructions, questionnaires and protocol-stated restrictions

Exclusion Criteria:

* Pregnant or lactating female
* Unstable patient who developed an exacerbation during the last 8 weeks
* Patient with upper or lower airways infection
* Patient unable to carry out pulmonary function testing
* Patient with an uncontrolled disease or any condition that might, in the judgement of the investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study
* Patient with cancer or any other chronic disease with poor prognosis and /or affecting patient status
* Patient with allergy, sensitivity or intolerance to study drugs and/or study drug formulation ingredients
* Patient unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study
* Patient who received oral corticosteroids within the last 4 weeks prior to visit 1
* Patient who received any investigational new drug within the last 4 weeks prior to visit 1 or twice the duration of the biological effect of any drug (whichever is longer)
* Patient with a history of alcohol or substance abuse that in the opinion of the investigator may be of clinical significance
* Patient who has undergone major surgery in the last 12 weeks before the visit 1 or has planned to undergo a major surgery before the end of the trial
* Patient with diagnosis of chronic obstructive pulmonary disease (COPD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Total airway volume | At visit 2 (= 7-11 days after visit 1)
  The primary objective of this study is to evaluate the effect of both the study drugs under investigation on Functional Respiratory Imaging (FRI) parameters and to evaluate the particle deposition in the lungs using Computational Fluid Dynamic (CFD)
The number of deposited particles per pre-defined airway section | At visit 2 (= 7-11 days after visit 1)
  The primary objective of this study is to evaluate the effect of both the study drugs under investigation on Functional Respiratory Imaging (FRI) parameters and to evaluate the particle deposition in the lungs using Computational Fluid Dynamic (CFD)
Total airway resistance | At visit 2 (= 7-11 days after visit 1)
  The primary objective of this study is to evaluate the effect of both the study drugs under investigation on Functional Respiratory Imaging (FRI) parameters and to evaluate the particle deposition in the lungs using Computational Fluid Dynamic (CFD)
Total airway volume | At visit 3 (= 3-7 days after visit 2)
  The primary objective of this study is to evaluate the effect of both the study drugs under investigation on Functional Respiratory Imaging (FRI) parameters and to evaluate the particle deposition in the lungs using Computational Fluid Dynamic (CFD)
The number of deposited particles per pre-defined airway section | At visit 3 (= 3-7 days after visit 2)
  The primary objective of this study is to evaluate the effect of both the study drugs under investigation on Functional Respiratory Imaging (FRI) parameters and to evaluate the particle deposition in the lungs using Computational Fluid Dynamic (CFD)
Total airway resistance | At visit 3 (= 3-7 days after visit 2)
  The primary objective of this study is to evaluate the effect of both the study drugs under investigation on Functional Respiratory Imaging (FRI) parameters and to evaluate the particle deposition in the lungs using Computational Fluid Dynamic (CFD)

SECONDARY OUTCOMES:
Lung function tests (spirometry, body plethysmography) | At visit 2 (= 7-11 days after visit 1)
  The secondary objectives are to assess the effect of both the study drugs on lung function (spirometry and body plethysmography), on exercise capacity (6 Minutes Walking Test = 6MWT) and on dyspnea (Borg Category (C) Ratio (R) 10 Scale and Visual Analog Scale (VAS) dyspnea).
Exercise capacity (6 minutes walking test) | At visit 2 (= 7-11 days after visit 1)
  The secondary objectives are to assess the effect of both the study drugs on lung function (spirometry and body plethysmography), on exercise capacity (6 Minutes Walking Test = 6MWT) and on dyspnea (Borg Category (C) Ratio (R) 10 Scale and Visual Analog Scale (VAS) dyspnea).
Dyspnea (BORG CR 10 scale and VAS dyspnea) | At visit 2 (= 7-11 days after visit 1)
  The secondary objectives are to assess the effect of both the study drugs on lung function (spirometry and body plethysmography), on exercise capacity (6 Minutes Walking Test = 6MWT) and on dyspnea (Borg Category (C) Ratio (R) 10 Scale and Visual Analog Scale (VAS) dyspnea).
Incidence of adverse events | From visit 1 until visit 4 = timeperiod of 3 à 4 weeks
  The safety of the 2 products under investigation will be evaluated through monitoring of adverse events (AEs) throughout the study.
Lung function tests (spirometry, body plethysmography) | At visit 3 (= 3-7 days after visit 2)
  The secondary objectives are to assess the effect of both the study drugs on lung function (spirometry and body plethysmography), on exercise capacity (6 Minutes Walking Test = 6MWT) and on dyspnea (Borg Category (C) Ratio (R) 10 Scale and Visual Analog Scale (VAS) dyspnea).
Exercise capacity (6 minutes walking test) | At visit 3 (= 3-7 days after visit 2)
  The secondary objectives are to assess the effect of both the study drugs on lung function (spirometry and body plethysmography), on exercise capacity (6 Minutes Walking Test = 6MWT) and on dyspnea (Borg Category (C) Ratio (R) 10 Scale and Visual Analog Scale (VAS) dyspnea).
Dyspnea (BORG CR 10 scale and VAS dyspnea) | At visit 3 (= 3-7 days after visit 2)
  The secondary objectives are to assess the effect of both the study drugs on lung function (spirometry and body plethysmography), on exercise capacity (6 Minutes Walking Test = 6MWT) and on dyspnea (Borg Category (C) Ratio (R) 10 Scale and Visual Analog Scale (VAS) dyspnea).

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

REFERENCES:
- [Derived] De Backer J, Van Holsbeke C, Vos W, Vinchurkar S, Dorinsky P, Rebello J, Mangale M, Hajian B, De Backer W. Assessment of lung deposition and analysis of the effect of fluticasone/salmeterol hydrofluoroalkane (HFA) pressurized metered dose inhaler (pMDI) in stable persistent asthma patients using functional respiratory imaging. Expert Rev Respir Med. 2016 Aug;10(8):927-33. doi: 10.1080/17476348.2016.1192464. Epub 2016 Jun 1. PMID 27227384